CLINICAL TRIAL: NCT04878627
Title: The Role of Cannabidiol in Regulating Meal Time Anxiety in Anorexia Nervous: Safety, Tolerability and Pharmacokinetics
Brief Title: Role of CBD in Regulating Meal Time Anxiety in Anorexia Nervosa
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Guido Frank, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191570
Record Dates: First submitted 2021-04-26; First posted 2021-05-07 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, randomized, double-blind study
Who Masked: Participant, Investigator
Masking Description: The PI and research coordinator administering the medication will be blinded to the randomization schedule. The research subject will be blinded to what medication she receives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cannabidiol (CBD) (Experimental): Days 1 to 7: Patients will receive CBD 2.5 mg/kg in divided doses BID for 7 days. Days 8 to 14: Patients will receive an increase dose of 7.5 mg/kg of CBD in divided doses.
  Days 15 to 21: Patients will receive an increased dose of 12.5 mg/kg CBD, in divided doses. If patients experience dose limiting side-effects, they ill be maintained on the lowest tolerated dose.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Days 1 to 7: Patients will receive placebo in divided doses BID for 7 days. Days 8 to 14: Patients will continue to receive placebo in divided doses. Days 15 to 21: Patients will receive continue to receive placebo in divided doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — patients receive cannabidiol at various doses for 3 weeks
  Other Names: Epidiolex
  Arms: Cannabidiol (CBD)
Drug: Placebo — patients receive placebo for 3 weeks
  Arms: Placebo

SUMMARY:
No studies of cannabidiol (CBD) have focused on Anorexia Nervosa (AN). Dose, side effects, tolerability, acceptability of pure CBD in AN must be established. The current study is an important first step in the investigation of CBD for AN. Cannabis products have been recently legalized in many states, and CBD in particular has been shown to reduce anxiety. Therefore, CBD may represent a promising new treatment for AN. The endocannabinoid system is involved in the regulation of functions relevant to eating disorders. Furthermore, data suggest that eating disorders are associated with alterations of the endocannabinoid system. Prior attempts to target the endocannabinoid system in AN have focused on CB1 receptor agonists that can increase anxiety. Moreover, CBD may be particularly beneficial in decreasing anxiety in AN via its action at serotonin receptors. Lastly, the impact of CBD on eating behavior and weight in AN must be determined. The current study seeks to explore these hypotheses using the aims in the following section.

ELIGIBILITY:
Inclusion Criteria:

1. Must currently meet DSM-5 criteria for AN-R and AN Spectrum Disorders (i.e., Atypical AN) based on the Structured Clinical Interview for the DSM-5 (SCID-5-RV)
2. Have a duration of illness ≥ 6 months
3. Be medically stable as assessed by a comprehensive medical and behavioral evaluation conducted by a study physician

Exclusion Criteria:

1. Psychotic illness/other mental illness requiring inpatient hospitalization
2. Current dependence on drugs or alcohol
3. Physical conditions (e.g., diabetes mellitus, pregnancy) known to influence eating or weight or liver disease which may affect pharmacokinetics of the study drug
4. Use of other psychoactive medications
5. Significant changes in medication in past month
6. Expression of acute suicidality
7. Previous hypersensitivity reaction to Epidiolex or any of its constituents

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female individuals will be enrolled. Gender eligibility is based on biological sex of participants.
Enrollment: 40 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Committee of Clinical Investigations UKU-Side Effect Scale Week 1 | After completion of Week 1 of treatment
  The Committee of Clinical Investigations (UKU) scale is used to rate psychiatric (e.g., depression, failing memory, concentration difficulty), neurological (e.g., rigidity, tremor, epileptic seizure), and autonomic (e.g., nausea, diarrhea, tachycardia) side effects, plus others. Higher scores indicate more side effects.
Committee of Clinical Investigations UKU-Side Effect Scale Week 2 | After completion of Week 2 of treatment
  The Committee of Clinical Investigations (UKU) scale is used to rate psychiatric (e.g., depression, failing memory, concentration difficulty), neurological (e.g., rigidity, tremor, epileptic seizure), and autonomic (e.g., nausea, diarrhea, tachycardia) side effects, plus others. Higher scores indicate more side effects.
Committee of Clinical Investigations UKU-Side Effect Scale Week 3 | After completion of Week 3 of treatment
  The Committee of Clinical Investigations (UKU) scale is used to rate psychiatric (e.g., depression, failing memory, concentration difficulty), neurological (e.g., rigidity, tremor, epileptic seizure), and autonomic (e.g., nausea, diarrhea, tachycardia) side effects, plus others. Higher scores indicate more side effects.
Blood tests for cannabinol (CBD) metabolites Week 1 | After Completion of Week 1 of treatment
  Blood levels for CBD, 6-OH-CBD, 7COOH-CBD, THC. The results will be compared to standard laboratory values.
Blood tests for cannabinol (CBD) metabolites Week 2 | After completion of Week 2 of treatment
  Blood levels for CBD, 6-OH-CBD, 7COOH-CBD, THC. The results will be compared to standard laboratory values.
Blood tests for cannabinol (CBD) metabolites Week 3 | After completion of Week 3 of treatment
  Blood levels for CBD, 6-OH-CBD, 7COOH-CBD, THC. The results will be compared to standard laboratory values.
Change from baseline scores of Eating Disorder Examination Questionnaire (EDE-Q) over the course of treatment | Weekly for the duration of the project (three weeks)
  Assesses the change from baseline in BMI, Eating Restraint, Eating Concern, Shape Concern, Weight Concern over the course of treatment. Each of those subscales is rated between 0 and 5. Subscales are calculated based on the average scores for the respective subscale. Higher scores indicate poorer outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Guido K Frank, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaye WH, Bulik CM, Thornton L, Barbarich N, Masters K. Comorbidity of anxiety disorders with anorexia and bulimia nervosa. Am J Psychiatry. 2004 Dec;161(12):2215-21. doi: 10.1176/appi.ajp.161.12.2215. PMID 15569892
- [Background] Ando T, Tamura N, Mera T, Morita C, Takei M, Nakamoto C, Koide M, Hotta M, Naruo T, Kawai K, Nakahara T, Yamaguchi C, Nagata T, Ookuma K, Okamoto Y, Yamanaka T, Kiriike N, Ichimaru Y, Ishikawa T, Komaki G; Japanese Genetic Research Group For Eating Disorders. Association of the c.385C>A (p.Pro129Thr) polymorphism of the fatty acid amide hydrolase gene with anorexia nervosa in the Japanese population. Mol Genet Genomic Med. 2014 Jul;2(4):313-8. doi: 10.1002/mgg3.69. Epub 2014 Feb 24. PMID 25077173
- [Background] Tambaro S, Bortolato M. Cannabinoid-related agents in the treatment of anxiety disorders: current knowledge and future perspectives. Recent Pat CNS Drug Discov. 2012 Apr 1;7(1):25-40. doi: 10.2174/157488912798842269. PMID 22280339
- [Background] Rong C, Lee Y, Carmona NE, Cha DS, Ragguett RM, Rosenblat JD, Mansur RB, Ho RC, McIntyre RS. Cannabidiol in medical marijuana: Research vistas and potential opportunities. Pharmacol Res. 2017 Jul;121:213-218. doi: 10.1016/j.phrs.2017.05.005. Epub 2017 May 10. PMID 28501518
- [Background] Bisogno T, Hanus L, De Petrocellis L, Tchilibon S, Ponde DE, Brandi I, Moriello AS, Davis JB, Mechoulam R, Di Marzo V. Molecular targets for cannabidiol and its synthetic analogues: effect on vanilloid VR1 receptors and on the cellular uptake and enzymatic hydrolysis of anandamide. Br J Pharmacol. 2001 Oct;134(4):845-52. doi: 10.1038/sj.bjp.0704327. PMID 11606325